CLINICAL TRIAL: NCT01427426
Title: Does a Nutritional Supplement Increase Vitality, Energy and Perceived Well Being?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Factors Group of Nutritional Companies Inc. (Industry); QualityMetrics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: H11-00426
Record Dates: First submitted 2011-08-05; First posted 2011-09-01 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Health; Vitality; Well-being; Nutritional Supplement; Phytonutrient; Greens

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- All Greens (Experimental): Subjects will consume the All Greens product daily. Product is prepared by mixing with either water, juice or in a smoothie.
  Interventions: Dietary Supplement: All Greens
- Control formulation (Sham Comparator): Subjects will consume a product of similar consistency and comparable taste that does not have the same healthy ingredients as the All Greens.
  Interventions: Other: Control Formulation

INTERVENTIONS:
Dietary Supplement: All Greens — All Greens is a mixture of organic alfalfa powder, barley, wheat grass juice powder, lycopene, cranberry juice extract, rosehips, grapeseed phytosomes, soya extract, Acidophilus, bromelain, apple pectin, and other ingredients. All Greens is approved by Health Canada and available to the public for purchase.
  Arms: All Greens
Other: Control Formulation — The Control Formulation is a rice-flour based product that has been designed to mimic the All Greens in appearance and taste.
  Arms: Control formulation

SUMMARY:
Factors Group is a producer of nutritional supplements. This study aims to determine whether one of their products improves the energy and sense of well-being in individuals who consume it. Interested subjects will complete a 1 week lead-in phase where they will be asked to consume a placebo daily to see if they are a good fit for the study. After the lead-in phase, subjects will be randomized to take either All Greens or a different placebo for 12 weeks. The investigators expect All Greens to have better results than the placebo, but subjects will not know which supplement they are taking. The primary outcome is a score on a questionnaire of well being.

DETAILED DESCRIPTION:
PURPOSE To conduct a study to determine the potential benefits of All Greens.

HYPOTHESIS Our primary hypothesis is that a greater proportion of participants on All Greens will score higher on the subjective scores of vitality and energy, as measured by our validated survey, than those consuming the control formulation.

JUSTIFICATION All Greens is a mixture of organic alfalfa powder, barley, wheat grass juice powder, lycopene, cranberry juice extract, rosehips, grapeseed phytosomes, soya extract, Acidophilus, bromelain, apple pectin, and other ingredients. All Greens is a well-balanced phytonutrient formula that nourishes, energizes, cleanses and acts as a whole body tonic. Recently, Boon et al (2004) have published results demonstrating some clinical benefits of consuming Greens+, a product similar to All Greens. After 12 weeks, women randomized to consume Greens+ scored marginally higher on subjective scores on Vitality and significantly higher on Energy than those consuming a placebo group (Boon, 2004). However, limitations of this study such as incomplete blinding and a high drop-out rate limit the veracity of the findings.

OBJECTIVES To determine if 12 weeks of consumption of All Greens increases vitality, energy, and perception of well-being compared to consumption of a placebo in adult women and men (18-45 y).

RESEARCH METHOD The investigators aim to recruit 120 people (18-45 y) through advertisements and word of mouth. In a lead-in phase, subjects will be asked to consume an 'initiation drink' daily for a week. The purpose of this is to identify those subjects who are unlikely to complete the study so they can be excluded before randomization, in order to minimize the dropout rate. The lead-in product will be composed primarily of rice flour, with other ingredients added to make it comparable to the All Greens and control formulation.

Participants remaining after the week lead-in phase week will be asked to attend a morning clinic at the university. Height and weight will be recorded, health and demographic information will be collected by questionnaire, and outcome measure questionnaires will be completed. Participants will be randomized to All Greens or the control formulation. Subjects will be instructed to record any side effects or adverse events in a study diary. At 6 weeks, study staff will phone participants, to check on progress.

Twelve weeks after randomization, participants will be asked to return to clinic to repeat the outcome measure questionnaires. Compliance will be assessed by weighing returned supplements and by patient diary. Adverse events will be recorded in the diaries. If patients withdraw from the study they will still be encouraged to return at 12 weeks to complete the outcome measures to allow for intent-to-treat analysis.

SAMPLE SIZE The sample size estimate is based on the primary outcome. The mean score on the vitality subscale of the SF-36 in a large study of women was 65 with a SD of 18. A ten-point change in the SF-36 vitality sub-scale can be considered a "moderate" effect that is clinically and socially relevant. Assuming 80% power, P-value of 0.05, an SD of 18, a correlation between baseline and follow-up measures of at least R=0.5, 50 subjects per treatment group would be needed to detect a 5 point difference between the groups. Assuming 20% attrition 120 subjects randomized would be required.

STATISTICAL ANALYSIS Differences in outcomes measures at twelve weeks will be assessed by multiple regression analysis with adjustment for baseline values and other predetermined factors (i.e. last menstrual period, oral contraceptive use).

ELIGIBILITY:
Inclusion Criteria:

* Not taking any other nutritional supplement (including fish oils, vitamins...) or be willing to discontinue use for duration of study

Exclusion Criteria:

* Medical conditions such as diabetes, asthma, cancer, cardiovascular disease, high blood pressure, celiac disease, a history of kidney stones or psychiatric illness.
* Currently taking antidepressants, anticoagulant or other medications that may interact with the nutritional supplement.
* Unable to provide informed consent
* Women who are pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in score on the Short-Form 36 (SF-36) | Baseline and Study End (12 weeks after randomization)
  The Short Form-36 (SF-36) is a validated, multi-purpose, short-form health survey that is a generic measure of health status/quality of life. It provides an overall measure of physical and mental health, as well as eight subscale profiles, of which three were considered to be relevant for this study: general health, vitality, and mental health. The SF-36 is licensed by the company QualityMetric.

SECONDARY OUTCOMES:
Change in scores on 10 cm Visual Analogue Scales (VAS) | Randomization and 12 weeks (study end)
  VAS scores will assess energy levels and sense of well being of subjects.
Number of participants who report side effects | From enrollment to 13 weeks (study end)
  Date, time, description, duration, frequency and severity (on a 5 point scale), of side effects will be recorded by the participant by use of a study diary.
Number of unused supplement packets | Enrollment to 13 weeks (study end)
  Compliance will be assessed by counting returned supplement packets as well as by review of the subject's study diary.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Green, PhD, Principal Investigator — University of British Columbia, Department of Food, Nutrition and Health
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Boon H, Clitheroe J, Forte T. Effects of greens+: a randomized, controlled trial. Can J Diet Pract Res. 2004 Summer;65(2):66-71. doi: 10.3148/65.2.2004.66. PMID 15217524